CLINICAL TRIAL: NCT04533685
Title: Patient Portal Reminder/Recall for Influenza Vaccination in a Health System- RCT 3
Brief Title: Patient Portal Reminder/Recall for Influenza Vaccination in a Health System- UCLA Portal R/R Influenza RCT 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-AM-00012; R01AI135029 (NIH)
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Vaccination; Reminder recall; Patient Portal
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: A 2x2x2 factorial design, nested within a parallel 2-arm trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Direct scheduling + Pre-commitment + Pre-appt reminder (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal with a link enabling direct scheduling, 2) a pre-commitment prompt and 3) pre-appointment reminders that mention asking the provider for a flu vaccine
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Direct scheduling link; Behavioral: Pre-Commitment Prompt; Behavioral: Pre-Appointment flu vaccine reminders
- Direct scheduling + Pre-commitment (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal with a link enabling direct scheduling and 2) a pre-commitment prompt
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Direct scheduling link; Behavioral: Pre-Commitment Prompt
- Direct scheduling + Pre-appt reminder (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal with a link enabling direct scheduling and 2) pre-appointment reminders that mention asking the provider for a flu vaccine
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Direct scheduling link; Behavioral: Pre-Appointment flu vaccine reminders
- Direct scheduling (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal with a link enabling direct scheduling
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: Direct scheduling link
- No direct scheduling + Pre-commitment + Pre-Appt reminder (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal without a link enabling direct scheduling, 2) a pre-commitment prompt and 3) pre-appointment reminders that mention asking the provider for a flu vaccine
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: No direct scheduling link; Behavioral: Pre-Commitment Prompt; Behavioral: Pre-Appointment flu vaccine reminders
- No direct scheduling + Pre-commitment (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal without a link enabling direct scheduling and 2) a pre-commitment prompt
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: No direct scheduling link; Behavioral: Pre-Commitment Prompt
- No direct scheduling + Pre-appt reminder (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal without a link enabling direct scheduling and 2) pre-appointment reminders that mention asking the provider for a flu vaccine
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: No direct scheduling link; Behavioral: Pre-Appointment flu vaccine reminders
- No direct scheduling (Active Comparator): Participants receive 1) reminder/recall messages regarding influenza vaccination via the patient portal without a link enabling direct scheduling for a flu vaccine appointment
  Interventions: Behavioral: Portal Reminders for Influenza Vaccination: No direct scheduling link
- Control Arm (No Intervention): Participants will not receive any reminder/recall messages regarding influenza vaccination via the patient portal or other intervention components

INTERVENTIONS:
Behavioral: Portal Reminders for Influenza Vaccination: Direct scheduling link — Patients receive reminder/recall messages via the patient portal to get an influenza vaccination that include a direct scheduling link, enabling the patient to directly schedule a flu vaccination only visit
  Arms: Direct scheduling; Direct scheduling + Pre-appt reminder; Direct scheduling + Pre-commitment; Direct scheduling + Pre-commitment + Pre-appt reminder
Behavioral: Portal Reminders for Influenza Vaccination: No direct scheduling link — Patients receive reminder/recall messages via the patient portal to get an influenza vaccination (no direct scheduling link included)
  Arms: No direct scheduling; No direct scheduling + Pre-appt reminder; No direct scheduling + Pre-commitment; No direct scheduling + Pre-commitment + Pre-Appt reminder
Behavioral: Pre-Commitment Prompt — Patients receive a pre-commitment prompt asking about their intention to get an influenza vaccination
  Arms: Direct scheduling + Pre-commitment; Direct scheduling + Pre-commitment + Pre-appt reminder; No direct scheduling + Pre-commitment; No direct scheduling + Pre-commitment + Pre-Appt reminder
Behavioral: Pre-Appointment flu vaccine reminders — Patients receive modified pre-appointment reminders for upcoming scheduled appointments that include language encouraging patients to ask the provider for the flu vaccine
  Arms: Direct scheduling + Pre-appt reminder; Direct scheduling + Pre-commitment + Pre-appt reminder; No direct scheduling + Pre-appt reminder; No direct scheduling + Pre-commitment + Pre-Appt reminder

SUMMARY:
This trial is taking place in Los Angeles, CA among patients from primary care practices within the UCLA Health System.

The study design is a 2x2x2 factorial design, nested in a parallel 2-arm trial. The parallel arms are control v. reminder letter (reminder messages sent via the patient portal, reminding participants of an overdue influenza vaccine)

Nested within the reminder letter arm, we will have 3 additional components:

* A direct scheduling link within the reminder letter enabling the patient to schedule an influenza vaccine only visit (direct scheduling link vs. no direct scheduling link).
* A pre-commitment prompt (pre-commitment prompt vs. no prompt) asking about a patient's intention to get the influenza vaccination
* A pre-appointment reminder, encouraging patients to ask for their influenza vaccine at their upcoming appointment (pre-appointment reminder encouraging influenza vaccination vs. standard pre-appointment reminder not mentioning influenza vaccination)

DETAILED DESCRIPTION:
This trial is taking place in Los Angeles, CA among patients from primary care practices within the UCLA Health System, using 2x2x2 factorial design, nested in a parallel 2-arm trial.

Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. For influenza specifically, annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Reminder/recall (R/R) messages, sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, the majority of pediatric or adult primary care practices to not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients.

This randomized controlled trial will assess the effectiveness of reminders messages, encouraging influenza vaccination, sent to patient portal users on increasing influenza vaccination rates within a health system by randomizing patients to two groups: 1) two-thirds of patients will receive reminder letters, 2) one-third will not receive reminders.

Patients in the reminder arm will be further randomized (separately) for three additional components: 1) direct appointment scheduling, 2) pre-commitment prompts and 3) pre-appointment reminders.

Direct scheduling: The convenience of scheduling an appointment for influenza vaccination may increase the likelihood that patients receive an influenza vaccination. Patients receiving reminders will be randomized to receive one of two types of reminder letters: 1) one half will receive flu vaccine reminder letters with a link to the MyChart direct appointment scheduling page and 2) one half will receive flu vaccine reminder message without the direct appointment scheduling link.

Pre-commitment: Another potential influence on the decision to vaccinate is pre-commitment. Previous studies suggest that, upon being prompted, indicating an intention to do something increases the likelihood of following through. Patients will be randomized to one of two groups: 1) one half will receive pre-commitment prompt at the beginning of influenza vaccination season and 2) one half will not receive a pre-commitment prompt. The pre-commitment prompt asks whether the patient intends to receive influenza vaccine, and where and when they plan to get the vaccine.

Pre-appointment flu reminders: Finally, a missed opportunities for vaccination occurs when patients are eligible for vaccination but are not offered a vaccine at their medical appointment. Pre-appointment reminders, sent in advance of an upcoming appointment, encouraging the patient talk to their doctor about influenza vaccination, may increase the likelihood of that patient receiving a vaccine. Patients will be randomized to one of two groups: 1) one half will receive modified pre-appointment reminders that mention influenza vaccination and 2) one half will receive the standard pre-appointment reminders for an upcoming appointment (no mention of influenza vaccination).

ELIGIBILITY:
Inclusion Criteria:

A patient within the UCLA Health System identified as a primary care patient per an internal algorithm.

Exclusion Criteria:

A patient within the UCLA Health System not identified as a primary care patient per an internal algorithm

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 213773 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Szilagyi, MD, MPH, Principal Investigator — Professor of Pediatrics
Locations (1):
- University of California LA, Los Angeles, California, United States

REFERENCES:
- [Derived] Szilagyi PG, Casillas A, Duru OK, Ong MK, Vangala S, Tseng CH, Albertin C, Humiston SG, Ross MK, Friedman SR, Evans S, Sloyan M, Bogard JE, Fox CR, Lerner C. Evaluation of behavioral economic strategies to raise influenza vaccination rates across a health system: Results from a randomized clinical trial. Prev Med. 2023 May;170:107474. doi: 10.1016/j.ypmed.2023.107474. Epub 2023 Mar 2. PMID 36870572

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct Scheduling + Pre-commitment + Pre-appt Reminder | Direct Scheduling + Pre-commitment | Direct Scheduling + Pre-appt Reminder | Direct Scheduling | No Direct Scheduling + Pre-commitment + Pre-Appt Reminder | No Direct Scheduling + Pre-commitment | No Direct Scheduling + Pre-appt Reminder | No Direct Scheduling | Control Arm
Started | 17848 | 17842 | 17832 | 17827 | 17821 | 17819 | 17812 | 17805 | 71167
Completed | 17848 | 17842 | 17832 | 17827 | 17821 | 17819 | 17812 | 17805 | 71167
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Scheduling + Pre-commitment + Pre-appt Reminder | Direct Scheduling + Pre-commitment | Direct Scheduling + Pre-appt Reminder | Direct Scheduling | No Direct Scheduling + Pre-commitment + Pre-Appt Reminder | No Direct Scheduling + Pre-commitment | No Direct Scheduling + Pre-appt Reminder | No Direct Scheduling | Control Arm | Total
Number analyzed (Participants) | 17848 | 17842 | 17832 | 17827 | 17821 | 17819 | 17812 | 17805 | 71167 | 213773
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 1556 | 1561 | 1535 | 1547 | 1511 | 1535 | 1546 | 1576 | 6071 | 18438
  18-64 years | 13166 | 13234 | 13208 | 13202 | 13274 | 13148 | 13238 | 13122 | 52973 | 158565
  65+ years | 3126 | 3047 | 3089 | 3078 | 3036 | 3136 | 3028 | 3107 | 12123 | 36770
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10100 | 10130 | 10158 | 10028 | 10179 | 10169 | 10116 | 10190 | 40517 | 121587
  Male | 7748 | 7711 | 7674 | 7797 | 7642 | 7648 | 7696 | 7615 | 30646 | 92177
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 9705 | 9501 | 9662 | 9676 | 9557 | 9648 | 9602 | 9628 | 38560 | 115539
  Asian | 1638 | 1756 | 1713 | 1703 | 1713 | 1793 | 1677 | 1770 | 6750 | 20513
  Black | 826 | 814 | 821 | 849 | 837 | 811 | 787 | 829 | 3332 | 9906
  American Indian or Alaska Native | 49 | 53 | 43 | 46 | 43 | 34 | 41 | 47 | 127 | 483
  Multiracial | 526 | 527 | 500 | 517 | 522 | 539 | 476 | 494 | 2022 | 6123
  Other | 2449 | 2491 | 2456 | 2472 | 2475 | 2439 | 2509 | 2465 | 9796 | 29552
  Unknown | 2620 | 2677 | 2597 | 2534 | 2637 | 2528 | 2686 | 2540 | 10406 | 31225
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 13227 | 13081 | 13272 | 13271 | 13164 | 13235 | 13111 | 13221 | 52663 | 158245
  Hispanic or Latino | 1802 | 1840 | 1828 | 1877 | 1894 | 1857 | 1883 | 1868 | 7400 | 22249
  Unknown | 2819 | 2921 | 2732 | 2679 | 2763 | 2727 | 2818 | 2716 | 11104 | 33279
Primary Language [Count of Participants; unit: Participants]
  English | 17504 | 17518 | 17521 | 17522 | 17451 | 17420 | 17451 | 17448 | 69771 | 209606
  Spanish | 134 | 133 | 135 | 122 | 130 | 157 | 145 | 155 | 525 | 1636
  Other | 192 | 180 | 166 | 171 | 231 | 227 | 198 | 188 | 800 | 2353
  Uknown | 18 | 11 | 10 | 12 | 9 | 15 | 18 | 14 | 71 | 178
Primary Insurance Class [Count of Participants; unit: Participants]
  Commercial | 12407 | 12544 | 12458 | 12393 | 12562 | 12443 | 12581 | 12367 | 49916 | 149671
  UCLA Managed Care | 2688 | 2700 | 2662 | 2760 | 2648 | 2683 | 2623 | 2723 | 10566 | 32053
  Medicare | 2055 | 1938 | 2040 | 2025 | 1950 | 2023 | 1967 | 2043 | 7949 | 23990
  Medi-Cal | 280 | 261 | 270 | 260 | 247 | 265 | 263 | 242 | 1063 | 3151
  Other | 223 | 216 | 217 | 195 | 220 | 197 | 190 | 226 | 888 | 2572
  Tricare | 108 | 106 | 123 | 121 | 125 | 120 | 109 | 117 | 475 | 1404
  Group Health Plan | 42 | 38 | 27 | 37 | 36 | 49 | 31 | 42 | 160 | 462
  International Payor | 5 | 4 | 3 | 3 | 4 | 5 | 6 | 5 | 12 | 47
  Self-pay | 3 | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 5 | 20
  Package Billing | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 5
  Unknown | 36 | 33 | 30 | 31 | 28 | 31 | 40 | 36 | 133 | 398

OUTCOME MEASURES:

1. Primary Outcome: Number of Index Patients Who Received Annual Influenza Vaccine
Description: Receipt of the annual influenza vaccination (between 8/1/20 - 4/1/21) among index patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data.
  The index patients must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 8/1/20, excluding activity on the user's initial profile activation date). Individuals not affiliated with any primary care practice will be excluded from the primary analysis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Scheduling + Pre-commitment + Pre-appt Reminder | Direct Scheduling + Pre-commitment | Direct Scheduling + Pre-appt Reminder | Direct Scheduling | No Direct Scheduling + Pre-commitment + Pre-Appt Reminder | No Direct Scheduling + Pre-commitment | No Direct Scheduling + Pre-appt Reminder | No Direct Scheduling | Control Arm
Number analyzed (Participants) | 17848 | 17842 | 17832 | 17827 | 17821 | 17819 | 17812 | 17805 | 71167
Participants | 6982 | 6988 | 6920 | 6990 | 7002 | 6999 | 6945 | 6891 | 27645
Statistical Analysis 1: Comparison: Direct Scheduling + Pre-commitment + Pre-appt Reminder vs Direct Scheduling + Pre-commitment vs Direct Scheduling + Pre-appt Reminder vs Direct Scheduling vs No Direct Scheduling + Pre-commitment + Pre-Appt Reminder vs No Direct Scheduling + Pre-commitment vs No Direct Scheduling + Pre-appt Reminder vs No Direct Scheduling; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.01, 95% CI 2-sided [1.00 to 1.02] — Adjusted risk ratio. These results compare arms which received reminder letters to the arm receiving no reminder letter (control)
Statistical Analysis 2: Comparison: Direct Scheduling + Pre-commitment + Pre-appt Reminder vs Direct Scheduling + Pre-commitment vs Direct Scheduling + Pre-appt Reminder vs Direct Scheduling vs No Direct Scheduling + Pre-commitment + Pre-Appt Reminder vs No Direct Scheduling + Pre-commitment vs No Direct Scheduling + Pre-appt Reminder vs No Direct Scheduling; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.00, 95% CI 2-sided [0.98 to 1.01] — These results compare arms which received direct appointment scheduling to the arms not receiving direct appointment scheduling
Statistical Analysis 3: Comparison: Direct Scheduling + Pre-commitment + Pre-appt Reminder vs Direct Scheduling + Pre-commitment vs Direct Scheduling + Pre-appt Reminder vs Direct Scheduling vs No Direct Scheduling + Pre-commitment + Pre-Appt Reminder vs No Direct Scheduling + Pre-commitment vs No Direct Scheduling + Pre-appt Reminder vs No Direct Scheduling; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.00, 95% CI 2-sided [1.00 to 1.01] — These results compare arms which received pre-commitment reminders to the arms not receiving pre-commitment reminders
Statistical Analysis 4: Comparison: Direct Scheduling + Pre-commitment + Pre-appt Reminder vs Direct Scheduling + Pre-commitment vs Direct Scheduling + Pre-appt Reminder vs Direct Scheduling vs No Direct Scheduling + Pre-commitment + Pre-Appt Reminder vs No Direct Scheduling + Pre-commitment vs No Direct Scheduling + Pre-appt Reminder vs No Direct Scheduling; Comparing the risk of receiving an influenza vaccination; Test type: Superiority; Adjusted Risk Ratio = 1.00, 95% CI 2-sided [0.99 to 1.01] — These results compare arms which received pre-appointment reminder to the arms not receiving pre-appointment reminder

ADVERSE EVENTS:
Time Frame: We did not collect information regarding adverse events.
Description: We did not collect adverse event information. We monitored whether reminder recall through the portal was effective at increased influenza vaccination rates. Because influenza vaccination is recommended by the Advisory Committee on Immunization Practices and is part of the U.S. recommended vaccine schedule, we did not collect adverse event data.
Arm/Group | Direct Scheduling + Pre-commitment + Pre-appt Reminder | Direct Scheduling + Pre-commitment | Direct Scheduling + Pre-appt Reminder | Direct Scheduling | No Direct Scheduling + Pre-commitment + Pre-Appt Reminder | No Direct Scheduling + Pre-commitment | No Direct Scheduling + Pre-appt Reminder | No Direct Scheduling | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04533685/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04533685/SAP_001.pdf